CLINICAL TRIAL: NCT06640140
Title: Effects of a Supervised Training Program on Functional Capacity in Patients With Heart Failure and Cardiorenal Syndrome
Brief Title: Effects of a Supervised Training Program on Functional Capacity in Patients With HF and Cardiorenal Syndrome
Acronym: Train-CR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Train-CR
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure; Cardiorenal Syndrome
Keywords: Heart failure; Cardiorenal Syndrome; Functional Capacity
MeSH Terms: conditions — Heart Failure; Cardio-Renal Syndrome | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: This is a prospective study, blinded for the evaluator, randomized (1:1) to receive standard management alone or combined with a training program (aerobic combined with strength exercises) that will be carried out in a single center.
Who Masked: Investigator
Masking Description: Blinded only for the evaluator of primary and secondary endpoints.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Patients allocated to this arm will receive the usual care plus explicit recommendations for home-based aerobic and strength training.
- Supervised aerobic plus strenght training (Active Comparator): Patients allocated to this arm will receive the usual care plus supervised aerobic and strength training.
  Interventions: Behavioral: Supervised aerobic plus strength training

INTERVENTIONS:
Behavioral: Supervised aerobic plus strength training — Supervised moderate to high-intensity interval aerobic training plus moderate to high-intensity strength training.
  Arms: Supervised aerobic plus strenght training

SUMMARY:
This is a prospective study, blinded for the evaluator, randomized (1:1) to receive standard management alone or combined with a training program (aerobic combined with strength exercises) that will be carried out in a single center. After randomization, patients will be clinically evaluated. The primary endpoint (peakVO2) will be assessed by cardiopulmonary exercise testing combined with echocardiography (echo-CPET) at 12 weeks. Ambulatory patients with heart failure and cardiorenal syndrome and functional class NYHA II-III will be enrolled. A sample size estimation [alfa: 0.05, power: 80%, a 20% loss rate, and at least a delta change of mean peakVO2: +2,4 mL/kg/min (SD±2)] of 26 patients (13 per arm) would be necessary to test our hypothesis.

DETAILED DESCRIPTION:
Heart failure (HF) is a highly prevalent clinical entity that predominantly affects elderly people with comorbidities. Among these, chronic kidney disease is particularly frequent, complicating disease management and worsening prognosis. Supervised training programs in patients with HF have improved functional capacity and reduced hospitalizations. However, the evidence is scarce regarding the effects of a supervised training program on patients with HF and cardiorenal syndrome. This work aims to evaluate the effect of a supervised exercise program for 12 weeks in patients with HF and cardiorenal syndrome on peak oxygen consumption (peakVO2).

This is a prospective study, blinded for the evaluator, randomized (1:1) to receive standard management alone or combined with a training program (aerobic combined with strength exercises) that will be carried out in a single center. After randomization, patients will be clinically evaluated. The primary endpoint (peakVO2) will be assessed by cardiopulmonary exercise testing combined with echocardiography (echo-CPET) at 12 weeks. Ambulatory patients with heart failure and cardiorenal syndrome and functional class NYHA II-III will be enrolled. A sample size estimation [alfa: 0.05, power: 80%, a 20% loss rate, and at least a delta change of mean peakVO2: +2,4 mL/kg/min (SD±2)] of 26 patients (13 per arm) would be necessary to test our hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with heart failure according to 2021 ESC guidelines for Heart Failure.
* Evidence of cardiorenal syndrome, defined as coexistent very high risk chronic kidney disease (CKD) (estimated glomerular filtration rate [eGFR] <30 ml/min/1.73m2 or eGFR 30 to 44 ml/min/1.73m2 and Urine Albumin-Creatinine Ratio [uACR] >30 mg/g) or rapidly progressive CKD (loss of >5 ml/min/1.73m2 in one year).
* Stable symptomatic heart failure patients (New York Heart Association functional class II-III/IV) during the last month.
* Age ≥ 18 years old.
* Willing to provide written informed consent.

Exclusion Criteria:

* Inability to perform a valid baseline cardiopulmonary exercise test.
* Significant primary severe valve disease that is considered the main symptom driver.
* Effort angina or signs of ischemia during CPET.
* Primary cardiomyopathies.
* Cardiac transplantation.
* Any other comorbidity with a life expectancy of less than one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-10-08 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Peak oxygen consumption | The investigators will evaluate peak oxygen consumption at baseline (week 0) and at week 12.
  Primary outcome: changes in peak oxygen consumption between groups at 12 weeks.
  Description:
  Peak oxigen consumption (also known as maximal functional capacity) will be evaluated using incremental and symptom-limited cardiopulmonary exercise testing on a semi-supine bicycle ergometer (coupled with stress echocardiography), beginning with a workload of 10 Watts and increasing gradually in a ramp protocol at 10-Watts increments every 1 minute. Peak oxygen consumption (PeakVO2) is defined as the highest value of VO2 during the last 20 seconds of exercise.
  Unit of measure of peak oxygen consumption: mL/kg/min (this is a directly reported measure from the cardiopulmonary exercise testing, not an aggregated or derived calculation).

SECONDARY OUTCOMES:
Kansas City Cardiomyopathy Questionnaire | The investigators will evaluate Kansas City Cardiomyopathy Questionnaire at baseline (week 0) and at week 12.
  The Kansas City Cardiomyopathy Questionnaire includes 23 items that map to 7 domains: symptom frequency, symptom burden, symptom stability, physical limitations, social limitations, quality of life, and self-efficacy (the patient's understanding of how to manage their heart failure). All Kansas City Cardiomyopathy Questionnaire domains are scaled from 0 to 100, where scores represent health status as follows: 0 to 24, very poor to poor; 25 to 49, poor to fair; 50 to 74, fair to good; and 75 to 100, good to excellent. A change of 5 points is considered to be a small but clinically important change, whereas changes of 10 and 20 points are considered moderate-to-large and large-to-very-large clinical changes.
Chronotropic index | The investigators will evaluate chronotropic index at baseline (week 0) and at week 12.
  Secondary outcome: changes in chronotropic response between groups at 12 weeks. Description: Chronotropic index is an index calculated in a maximal cardiopulmonary exercise testing to assess heart rate response to exercise. The chronotropic index is evaluated by the following formula, including heart rate at peak effort, heart rate at rest and age. Chronotropic index: (peak heart rate-rest heart rate)/ [220-age-rest heart rate)]. The chronotropic index has no units of measure.

OTHER OUTCOMES:
Age | The investigators will evaluate age at baseline (week 0) and at week 12.
  Age at the moment of assessment that will be used to further calculate chronotropic index.
  Units: years.
Peak heart rate | The investigators will evaluate peak heart rate at baseline (week 0) and at week 12.
  Peak heart rate is defined as heart rate at the end of exercise of the maximal cardiopulmonary exercise testing and will be used to further calculate chronotropic index.
  Units: beats per minute.
Heart rate at rest | The investigators will evaluate heart rate at rest at baseline (week 0) and at week 12.
  Heart rate at rest is defined as heart rate at the beginning of the maximal cardiopulmonary exercise testing and will be used to further calculate chronotropic index.
  Units: beats per minute.

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Núñez Marín, MD, Principal Investigator — Instituto de investigación sanitaria INCLIVA
Locations (1):
- Instituto de investigación sanitaria INCLIVA, Valencia, Spain